CLINICAL TRIAL: NCT06557265
Title: A Phase 1/2 Study of NKX019, a CD19 Chimeric Antigen Receptor Natural Killer (CAR NK) Cell Therapy, in Subjects With Autoimmune Disease
Brief Title: A Phase 1/2 Study of NKX019 in Subjects With Autoimmune Disease (Ntrust-1)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nkarta, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKX019-102
Record Dates: First submitted 2024-07-10; First posted 2024-08-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Lupus Nephritis; Primary Membranous Nephropathy
Keywords: CD19; CAR; Allogeneic; NKX019; Interleukin 15; Cell Therapy; Immunotherapy; Adoptive cell therapy; Lupus Nephritis; Ntrust-1; LN; Primary Membranous Nephropathy; pMN
MeSH Terms: conditions — Lupus Nephritis | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NKX019 - CAR NK cell therapy (Experimental): Phase 1/2: NKX019 plus fludarabine and cyclophosphamide
  Interventions: Drug: NKX019; Drug: Fludarabine, Cyclophosphamide

INTERVENTIONS:
Drug: NKX019 — NKX019 is an investigational allogeneic CD19-Directed CAR NK
Drug: Fludarabine, Cyclophosphamide — For Lymphodepletion

SUMMARY:
This is an open-label, multi-center, non-randomized, Phase 1/2 study to determine the safety and tolerability of NKX019 (allogeneic CAR NK cells targeting CD19) in participants with active lupus nephritis (LN) or primary membranous nephropathy (pMN).

DETAILED DESCRIPTION:
Dose escalation of NKX019 will utilize a "3+3" design to determine the recommended dose(s) for enrolling additional participants across indications. The study will evaluate safety and tolerability, preliminary efficacy, pharmacokinetics, pharmacodynamics in participants with autoimmune diseases. Participants will receive a cycle consisting of lymphodepletion with fludarabine and cyclophosphamide (Flu/Cy), followed by three doses of NKX019. Participants who are cytopenic may receive a modified LD regimen of Cy alone.

ELIGIBILITY:
General Inclusion Criteria:

1. Age ≥18 and ≤70
2. Progression despite maximal tolerated doses of renin-angiotensin system (RAS) blockade agents
3. For participants taking chronic corticosteroids for management of the disease under study, the prednisone (or equivalent) dose must be ≤40 mg/day at 6 weeks prior to Screening and stable for ≥ 14 days before start of Screening
4. Negative SARS-CoV-2 test
5. For subjects on immunosuppressives or immunomodulators (other than corticosteroids), all doses must be stable for ≥ 4 weeks prior to Screening

LN-specific Inclusion Criteria:

1. Score of 10 or more points on the American College of Rheumatology (ACR) 2019 classification criteria for SLE
2. Active biopsy proven lupus nephritis Class III or Class IV with or without Class V using the 2018 International Society of Nephrology and Renal Pathology Society (ISN/RPS) criteria (Bajema 2018) as evidenced on kidney biopsy during screening or within 6 months before screening. For subjects with primarily Class III or Class IV LN, the biopsy must have at least mild to moderate activity score (≥4/24) and no more than moderate chronicity index (≤ 6/12) per NIH indices
3. Active renal disease as defined by urinary protein:creatinine ratio (UPCR) ≥ 1.5 g/g or proteinuria ≥1.5 g/day on a 24-hour collection and ≤ 7 g/day by either measure
4. Positive antinuclear antibodies (ANA) ≥ 1:80 OR anti-dsDNA OR anti-Smith (anti-Sm)
5. Refractory LN defined as having received ≥ 2 prior therapies for LN (immunosuppressant and corticosteroid/or immunomodulatory agent, and corticosteroid at therapeutic range for at least 90 days), and had an inadequate response to therapy despite being on a therapeutic dose for ≥ 90 days

pMN-specific Inclusion Criteria:

1. Evidence of pMN by renal biopsy during screening or within 6 months before screening
2. Active renal disease at screening defined by spot UPCR ≥ 3.5 g/g or proteinuria ≥ 3.5 g/day on a 24-hour collection
3. Positive anti-PLA2R antibodies
4. Refractory or intolerant to at least one induction therapy for pMN (immunosuppressant and corticosteroid or immunomodulatory agent and/corticosteroid) and defined as not achieving a complete remission after 180 days, or partial remission after 90 days

General Exclusion Criteria:

1. eGFR < 45 ml/min/1.73 m^2
2. Currently requiring renal dialysis or expected to require dialysis during the study period
3. Previous solid organ or hematopoietic cell transplant or planned transplant within study treatment period
4. Congenital or acquired immunodeficiency resulting in severe infection or those receiving chronic immunoglobulin replacement therapy
5. Liver disease or dysfunction, including cirrhosis and/or aspartate aminotransferase, alanine aminotransferase, or bilirubin ≥ 3 times the upper limit of normal
6. Pulmonary comorbidity including chronic obstructive pulmonary disease or asthma requiring daily oral steroids, resting hypoxemia (<92% oxygen saturation via pulse oximetry) on room air, or significant smoking history (i.e. >10 pack/year) with active pulmonary disease
7. White blood cell count < 3,000/mm^3; hemoglobin levels < 9 gm/dL absolute neutrophil count < 2,000/mm^3; platelet count < 100,000/mm^3
8. Major cardiac disease, abnormalities, or interventions as defined by, but not limited to:

   1. Uncontrolled angina or unstable life-threatening arrhythmias
   2. History of myocardial infarction within 12 weeks prior to the first dose of NKX019
   3. Any prior coronary artery bypass graft surgery
   4. ≥ Class III New York Heart Association (NYHA) congestive heart failure (CHF), significantly decreased ejection fraction (EF ≤ 40%), or severe cardiac insufficiency.
   5. Prolongation of the QT interval corrected for heart rate (QTc) (Fridericia) interval of > 480 msec
   6. Peripheral artery bypass graft surgery, pulmonary embolism, or other ≥ Grade 2 thrombotic or embolic events within 12 weeks prior to the first dose of NKX019
   7. Uncontrolled hypertension (systolic blood pressure > 160mmHg and diastolic > 90mmHg) despite therapy
9. Active bleeding disorders
10. Any overlapping autoimmune condition for which the condition itself or the treatment of that condition may affect the study assessments or outcomes; clinically significant conditions that could cause a secondary nephropathy; or kidney biopsy-confirmed significant renal disease other than disease under study
11. Pregnancy, breast feeding or, if of childbearing potential, not using adequate contraceptive precautions
12. Current infection requiring active systemic anti-infective therapy or recent acute infection requiring systemic therapy within 30 days of planned LD
13. History of positive HIV antibody or test positive at screening, Hepatitis B or C positive at screening, active tuberculosis (TB) or latent TB requiring suppressive therapy
14. Major surgery within 28 days prior to the first dose of NKX019
15. Malignancy within 5 years of screening, with the exception of basal and squamous cell carcinomas treated by complete excision. Subjects with cervical dysplasia that is cervical intraepithelial neoplasia but have been treated with conization or loop electrosurgical excision procedure and have had a normal repeat Papanicolaou test are allowed
16. Prior cellular therapy
17. Central nervous system (CNS) comorbidity or any autoimmune disease with CNS involvement within 90 days prior to the first dose of NKX019 as well as active CNS lupus within 1 year prior to screening
18. Any other acute or chronic medical or psychiatric condition, or known laboratory abnormality that, in the Investigator's opinion, is expected to interfere or impact study participation
19. Disease-modifying therapies for disease under study or investigational agents within 14 days or 5 half-lives of the drug (whichever is shorter), prior to LD.

    a. For those subjects on B-cell-depleting or -modulating drugs (ie, rituximab, belimumab), the subject must have received first dose ≥ 6 months prior to LD
20. Currently taking or known need for any of the medications prohibited in the study protocol
21. Known hypersensitivity or contraindications to the study treatment including LD; or other components such as human serum albumin or dimethyl sulfoxide

LN-specific Exclusion Criteria:

1. Known clinically active antiphospholipid antibody syndrome (APS); or high-risk profile

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From the first administration of NKX019 until the last administration of any study treatment + 30 days
  Incidence and severity of treatment-emergent adverse events will be evaluated
Incidence of dose-limiting toxicities (DLTs) [Safety and Tolerability] | The first 28 days after the first NKX019 dose
  Incidence of DLTs will be evaluated

SECONDARY OUTCOMES:
LN only: Number of participants who achieved Primary Efficacy Renal Response (PERR) (Furie 2020), complete renal response (CRR) and partial renal response (PRR) | Up to 2 years after NKX019 infusion
  Primary Efficacy Renal Response (PERR), complete renal response (CRR) and partial renal response (PRR) to treatment will be assessed based on European Alliance of Associations for Rheumatology (EULAR)/European Renal Association-European Dialysis and Transplantation Association (ERA-EDTA) criteria (Bertsias 2012)
LN only: Assessment of Lupus Low Disease Activity State (LLDAS) and Definition of Remission in SLE (DORIS) remission over time | Up to 2 years from NKX019 infusion
LN only: Change from baseline in Systemic Lupus Erythematosus (SLE) Disease Activity Index 2000 (SLEDAI-2K) score over time | Up to 2 years from NKX019 infusion
  The SLEDAI-2K score falls between 0 and 105. A higher score represents greater disease activity
pMN only: Number of participants who achieved complete remission (CR) and partial remission (PR) and their components (Couser 2017) | Up to 2 years from NKX019 infusion
pMN only: Change from baseline in serum albumin | Up to 2 years after NKX019 infusion
pMN only: % change from baseline in estimated glomerular filtration rate (eGFR) | Up to 2 years after NKX019 infusion
Maximum Concentration (Cmax) of NKX019 in peripheral blood | Up to 2 years after NKX019 infusion
Time to Cmax (Tmax) of NKX019 in peripheral blood | Up to 2 years after NKX019 infusion
Area Under the Concentration-time Curve (AUC) of NKX019 in peripheral blood | Up to 2 years after NKX019 infusion
Half-life (t1/2) of NKX019 in peripheral blood | Up to 2 years after NKX019 infusion
Duration of Persistence of NKX019 in peripheral blood | Up to 2 years after NKX019 infusion
Incidence of positive anti-NKX019 antibodies to assess immunogenicity of NKX019 over time | Up to 2 years after NKX019 infusion
Evaluation of the effect of treatment on background therapies | Up to 2 years after NKX019 infusion
  Proportion of subjects requiring rescue therapy over time
Evaluation of the effect of treatment on background therapies | Up to 2 years after NKX019 infusion
  Proportion of subjects who are steroid free over time
Evaluation of the effect of treatment on background therapies | Up to 2 years after NKX019 infusion
  Cumulative corticosteroid dose over time
Evaluation of the effect of treatment on background therapies | Up to 2 years after NKX019 infusion
  Proportion of subjects receiving ≤5 mg daily prednisone (or equivalent) over time
Evaluation of the effect of treatment on background therapies | Up to 2 years after NKX019 infusion
  Proportion of subjects receiving ≤7.5 mg daily prednisone (or equivalent) over time

CONTACTS AND LOCATIONS:
Overall Officials: Nkarta Study Director, Study Director — Nkarta, Inc.
Locations (15):
- United States (14):
  - Nkarta Investigational Site, Little Rock, Arkansas
  - Nkarta Investigational Site, Gainesville, Florida
  - Nkarta Investigational Site, Miami, Florida
  - Nkarta Investigational Site, Plantation, Florida
  - Nkarta Investigational Site, Atlanta, Georgia
  - Nkarta Investigational Site, Chicago, Illinois
  - Nkarta Investigational Site, New Orleans, Louisiana
  - Nkarta Investigational Site, Worcester, Massachusetts
  - Nkarta Investigational Site, Ann Arbor, Michigan
  - Nkarta Investigational Site, New York, New York
  - Nkarta Investigational Site, Stony Brook, New York
  - Nkarta Investigational Site, Syracuse, New York
  - Nkarta Investigational Site, Dallas, Texas
  - Nkarta Investigational Site, Houston, Texas
- Nkarta Investigational Site, Manatí, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Ntrust-1 Study for Lupus — https://www.ntrust1.com/